CLINICAL TRIAL: NCT02950584
Title: The Surface Roughness of Rapid Heat Cured Acrylic Resin Versus Modified Conventional Acrylic Resin With Titanium Dioxide Nanoparticles in Maxillary Single Dentures: A Randomized Clinical Trials
Brief Title: Surface Roughness of Heat Cured Acrylic Resin Versus Acrylic Resin With Titanium Dioxide
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, emad gamal ismail, Principal Investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 89
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Denture Stomatitis
MeSH Terms: conditions — Stomatitis, Denture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients take titanium dioxide denture (Experimental): Participants will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles) for 1 month in the initial phase of the trial then in the later phase after one month they will receive (rapid heat cured acrylic resin) denture
  Interventions: Other: Titanium dioxide denture; Other: Rapid heat denture
- Patients take rapid heat denture (Placebo Comparator): Patients will receive rapid heat denture for 1 month in the initial phase of the trial then in the later phase patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles)
  Interventions: Other: Titanium dioxide denture; Other: Rapid heat denture

INTERVENTIONS:
Other: Titanium dioxide denture — Patients will receive titanium dioxide denture (made from acrylic resin with titanium dioxide nanoparticles) for 1 month in the initial phase then in the second phase after one month they will receive (rapid heat cured acrylic resin)denture according to the principle of crossover design
Other: Rapid heat denture — Patients will receive rapid heat denture for 1 month in the initial phase of the trial then in the later phase patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles) according to the principle of crossover design

SUMMARY:
Measurement of surface roughness of tow different material of denture base to find out which material is more hygienic by decreasing the amount of bacterial accumulation.

DETAILED DESCRIPTION:
Using a denture base material as a standard value which is the rapid heat cured acrylic resin and compare it with a new material which is a conventional acrylic resin with addition of titanium dioxide nano particles in surface roughness and measuring it by a device called stylus profilometer this will be done on 20 patients this trial will take about 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous maxillary arch and fully dentate mandibular arch with adequate interarch space.
2. The edentulous ridges should be covered by firm healthy mucosa.
3. Angle class I maxillomandibular relationship
4. Healthy and co-operative patients

Exclusion Criteria:

1. Patients with bad habits as severe clenching or bruxism, drug or alcohol addiction, moderate or heavy smoking (greater than 10 cigarettes/day).
2. Previous history of radiotherapy or chemotherapy.
3. Any skeletal problem dictates surgical intervention

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The Surface Roughness of the denture base will be measured and reported in micrometer unit | 6 months
  surface profilometry will be measured by stylus profilometer

IPD SHARING:
Plan to Share IPD: Undecided